CLINICAL TRIAL: NCT06529523
Title: PD-1 (Programmed Cell Death Protein 1) Blockade in Mismatch-repair Deficient Colorectal Cancer in Nigeria
Brief Title: Tislelizumab in People With Colorectal Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: BeiGene USA, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 24-063
Record Dates: First submitted 2024-07-26; First posted 2024-07-31 (Actual); Last update posted 2025-10-07 (Actual); Status verified 2025-10

CONDITIONS: Colorectal Cancer
Keywords: Tislelizumab; PD-1 blockade; 24-063
MeSH Terms: conditions — Colorectal Neoplasms | interventions — tislelizumab

STUDY DESIGN:
Intervention Model Description: This is a pilot, open label to gather preliminary data on the use of PD-1 blockade therapy in patients with metastatic dMMR CRC (cohort 1) and patients with localized (stage II/III) dMMR rectal cancer (cohort 2).
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Cohort 1: Stage 4 Colorectal cancer (Experimental): All patients in the trial will be given Tislelizumab at a dose of 200mg IV over 30 minutes (60 minutes at the initial infusion), every 3 weeks.
  Interventions: Drug: Tislelizumab
- Cohort 2: Stage 2/3 Rectal cancer (Experimental): All patients in the trial will be given Tislelizumab at a dose of 200mg IV over 30 minutes (60 minutes at the initial infusion), every 3 weeks.
  Interventions: Drug: Tislelizumab

INTERVENTIONS:
Drug: Tislelizumab — Patients will receive standard dose of tislelizumab 200mg IV flat dose q3weeks until disease progression, unacceptable toxicity, patient/physician decides to withdraw patient, death, or completion of 104 weeks treatment (35 administrations).

SUMMARY:
The researchers are doing this study to find out whether tislelizumab is an effective treatment for people with colorectal cancer who are living in Nigeria. The researchers will also look at the safety of the study drug.

All participants in this study will be treatment naïve (they have not yet received treatment for their cancer), and their cancer will be mismatch repair deficient (dMMR). dMMR cancer can happen when your cells are unable to repair mistakes made during the cell division process.

ELIGIBILITY:
All subjects

Inclusion Criteria:

* Age 18 years or older on date of signing informed consent
* ECOG performance status of 0 or 1
* Negative pregnancy test done within 72 hours prior to start of treatment for women of childbearing potential.

  * Women of childbearing potential must be willing to use a highly effective method of birth control for the duration of the study and for ≥ 120 days after the last dose of tislelizumab They must also have a negative urine or serum pregnancy test result ≤ 7 days before first dose of study drug.
  * The Clinical Trials Facilitation Group recommendations related to contraception and pregnancy testing in clinical studies include the use of highly effective forms of birth control (Clinical Trials Facilitation Group 2014). These methods include the following:

    * Oral, intravaginal, or transdermal combined (estrogen- and progestogen-containing) hormonal contraception associated with the inhibition of ovulation
    * Oral, injectable, implantable progestogen-only hormonal contraception associated with the inhibition of ovulation Note: Oral birth control pills are not considered a highly effective form of birth control, and if they are selected, they must be used with a second, barrier method of contraception such as condoms with or without spermicide.
    * An intrauterine device
    * Intrauterine hormone-releasing system
    * Bilateral tubal occlusion
    * Vasectomized partner Note: This is only considered a highly effective form of birth control when the vasectomized partner is the sole partner of the study participant and there has been a medical assessment confirming surgical success.
    * A sterile male is one for whom azoospermia, in a semen sample, has been demonstrated as definitive evidence of infertility.
    * Sexual abstinence (defined as refraining from heterosexual intercourse during the entire period of risk associated with the study treatment) Note: Total sexual abstinence should only be used as a contraceptive method if it is in line with the patients' usual and preferred lifestyle.

Periodic abstinence (eg, calendar, ovulation, sympto-thermal, postovulation methods), declaration of abstinence for the duration of exposure to study drug, and withdrawal are not acceptable methods of contraception.

Of note, barrier contraception (including male and female condoms with or without spermicide) is not considered a highly effective method of contraception; if used, this method must be used in combination with one of the highly effective forms of birth control listed above.

°"Women of non-childbearing potential" are defined as female patients meeting any of the following criteria:

* Surgically sterile (ie, through bilateral salpingectomy, bilateral oophorectomy, or hysterectomy)
* Postmenopausal, defined as:

  * ≥ 55 years of age with no spontaneous menses for ≥ 12 months OR
  * < 55 years of age with no spontaneous menses for ≥ 12 months AND with postmenopausal follicle-stimulating hormone (FSH) concentration > 30 IU/mL and all alternative medical causes for the lack of spontaneous menses for ≥ 12 months have been ruled out, such as polycystic ovarian syndrome, hyperprolactinemia, etc.
  * If an FSH measurement is required to confirm postmenopausal state, concomitant use of hormonal contraception or hormonal replacement therapy should be excluded.

[Adapted from Clinical Trials Facilitation Group (CTFG) 2014.]

* Nonsterile males must be willing to use a highly effective method of birth control for the duration of the study and for ≥ 120 days after the last dose of tislelizumab

  •A sterile male is defined as one for whom azoospermia has been previously demonstrated in a semen sample examination as definitive evidence of infertility.
  * Males with known "low sperm counts" (consistent with "subfertility") are not to be considered sterile.

    - Demonstration of adequate organ function below within 14 days of cycle 1 day 1
    * The ability to adhere to the study protocol and willingness to provide informed consent
    * Cohort 1 subjects
  * Histological confirmation of colorectal adenocarcinoma
  * Confirmation of dMMR by immunohistochemistry
  * Radiologically measurable metastatic disease as per RECIST 1.1, not eligible for potentially curative surgery -Cohort 2 subjects
  * Histological confirmation of rectal adenocarcinoma
  * Confirmation of dMMR by immunohistochemistry
  * Rectal cancer stage II or III per AJCC 8 th edition criteria
  * No evidence of distant metastases

    * Hematological
* Absolute neutrophil count (ANC) ≥1,500 /mm^3
* Platelets ≥100,000 / mcL
* Hemoglobin >9 g/dL or ≥5.6 mmol/L

  * Renal
* Serum creatinine OR measured or calculated creatinine clearance (GFR can also be used in place of creatinine or CrCl) ≤1.5 × upper limit of normal (ULN) OR ≥30 mL/min for subject with creatinine levels > 1.5 × institutional ULN

  * Hepatic
* Serum total bilirubin ≤ 1.5 × ULN OR Direct bilirubin ≤ ULN for subjects with total bilirubin levels > 1.5 ULN
* AST (SGOT) and ALT (SGPT) ≤ 2.5 × ULN (< 5 x ULN if hepatic metastases are present in cohort 1

  * Coagulation
* International Normalized Ratio (INR) or Prothrombin Time (PT) Activated Partial Thromboplastin Time (aPTT) INR <1.5 or PT <1.5 x ULN; and either PTT or aPTT <1.5 x ULN. Patients on warfarin may be included on a stable dose with a therapeutic INR <3.5

Exclusion Criteria:

* Presence of other active malignancy
* Diagnosis of immunodeficiency or receiving systemic steroid therapy or other immunosuppressive therapy within 7 days prior to first dose of treatment
* Any condition that required systemic treatment with either corticosteroids (> 10 mg daily of prednisone or equivalent) or other immunosuppressive medication ≤ 14 days before first dose of study drug. Inhaled or topical steroids, and adrenal replacement doses > 10 mg daily prednisone equivalents are permitted in the absence of an active autoimmune disease. Note: Patients who are currently or have previously been on any of the following steroid regimens are not excluded:

  1. Adrenal replacement steroid (dose ≤ 10 mg daily of prednisone or equivalent)
  2. Topical, ocular, intra-articular, intranasal, or inhaled corticosteroid with minimal systemic absorption
  3. Short course (≤ 7 days) of corticosteroid prescribed prophylactically (eg, for contrast dye allergy) or for the treatment of a nonautoimmune condition (eg, delayed-type hypersensitivity reaction caused by contact allergen
* Active autoimmune disease requiring systemic therapy within the 2 years prior to treatment initiation

  o Well controlled hypothyroidism, diabetes, and skin conditions allowed
* Untreated active Hepatitis B or Hepatitis C

  o Patients actively on therapy with disease under control are allowed
* Untreated Acquired Immunodeficiency Syndrome (AIDS)

  o Patients with Human Immunodeficiency Virus (HIV) well controlled on anti-retroviral therapy are allowed
* Infection (including tuberculosis infection, etc.) requiring systemic (oral or intravenous) antibacterial, antifungal, or antiviral therapy ≤ 14 days before first dose of study drug
* History of interstitial lung disease, noninfectious pneumonitis, or uncontrolled lung diseases including pulmonary fibrosis.

  o Patients with significantly impaired pulmonary function or who require supplemental oxygen at baseline must undergo an assessment of pulmonary function at screening
* Currently receiving other anticancer or experimental therapy
* Has received prior therapy with an immune checkpoint inhibitor
* Prior ≥ Grade 3 immune-related AE from previous immunotherapy
* Pregnant women, women who are breast-feeding, or men expecting to conceive or father children during the trial period, through 120 days after last dose of medication
* Receipt of live vaccine within 30 days of planned treatment start
* Major surgical procedure or significant traumatic injury within 28 days prior to enrollment
* Known hypersensitivity to Tislelizumab
* Prior allogeneic stem cell or organ transplantation
* Any of the following cardiovascular risk factors:

  a. Cardiac chest pain, defined as moderate pain that limits instrumental activities of daily living, ≤ 28 days before first dose of study drug b. Pulmonary embolism ≤ 28 days before first dose of study drug c. Any history of acute myocardial infarction ≤ 6 months before first dose of study drug d. Any history of heart failure meeting New York Heart Association Classification III or IV ≤ 6 months before first dose of study drug e. Any event of ventricular arrhythmia ≥ Grade 2 in severity ≤ 6 months before first dose of study drug f. Any history of cerebrovascular accident ≤ 6 months before first dose of study drug g. Uncontrolled hypertension that cannot be managed by standard antihypertension medications ≤ 28 days before first dose of study drug h. Any episode of syncope or seizure ≤ 28 days before first dose of study drug
* Cohort 1 subjects
* Prior immunotherapy, chemotherapy, radiation therapy, or surgery for metastatic colorectal cancer

  o Treatment with adjuvant therapy of prior localized tumor is allowable as long as it was completed at least 6 months prior to cycle 1 day 1
* Known active central nervous system (CNS) metastasis and/or carcinomatous meningitis

  o Patients with previously treated brain metastases may participate if the brain metastases are stable via MRI assessment, performed ≥ 4 weeks after treatment
* Cohort 2 subjects
* Prior immunotherapy, chemotherapy, radiation therapy, or surgery for localized rectal cancer
* Presence of metastatic or recurrent disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-07-26 (Actual); Primary Completion 2028-07 (Estimated); Study Completion 2028-07 (Estimated)

PRIMARY OUTCOMES:
objective response rate of PD-1 blockade with tislelizumab | 2 years
  (ORR, defined as CR or PR) as measured by RECIST 1.1 in patients with mismatch repair deficient metastatic colorectal adenocarcinoma (cohort 1) and in patients with mismatch repair deficient localized (stage II/III) rectal adenocarcinoma (cohort 2).

CONTACTS AND LOCATIONS:
Overall Officials: Fiyinfolu O Balogun, MD, PhD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (3):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States
- Nigeria (2):
  - Lagos University Teaching Hospital, Idi Araba, Lagos
  - Obafemi Awolowo University Teaching Hospital, Ile-Ife

IPD SHARING:
Plan to Share IPD: Yes
Memorial Sloan Kettering Cancer Center supports the international committee of medical journal editors (ICMJE) and the ethical obligation of responsible sharing of data from clinical trials. The protocol summary, a statistical summary, and informed consent form will be made available on clinicaltrials.gov when required as a condition of Federal awards, other agreements supporting the research and/or as otherwise required. Requests for deidentified individual participant data can be made beginning 12 months after publication and for up to 36 months post publication. Deidentified individual participant data reported in the manuscript will be shared under the terms of a Data Use Agreement and may only be used for approved proposals. Requests may be made to: crdatashare@mskcc.org

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/mskcc/html/44.cfm